CLINICAL TRIAL: NCT05413707
Title: Posterior Malleolus Fractures (PMF) in Weber B Ankle Fractures - Fixation Versus no Fixation - a Randomized Controlled Trial
Brief Title: Weber B Ankle Fractures With Associated Posterior Malleolus Fracture
Acronym: PMFIX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: University Hospital, Akershus (Other); Ullevaal University Hospital (Other); Helse Stavanger HF (Other Government); Alesund Hospital (Other); Ostfold Hospital Trust (Other); St. Olavs Hospital (Other); Helgeland Hospital Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 255548
Record Dates: First submitted 2022-05-24; First posted 2022-06-10 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Posterior Malleolus Fractures; Ankle Fractures; Syndesmotic Injuries; Patient Reported Outcome Measure; Treatment Outcome
Keywords: Posterior malleolus fractures; Ankle factures; Weber B fractures; Syndesmotic injuries; Fixation; Randomized Controlled Trial
MeSH Terms: conditions — Ankle Fractures; Ankle Injuries

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with to arms: Fixation of posterior malleolus fractures (PMFs) versus no fixation of the PMF.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fixation group (Experimental): Patients are placed in a prone position on the operating table. Fixation of the posterior malleolus fracture. Posterior, and/or lateral and medial malleolus fractures will be treated with open reduction and internal fixation. ORIF of the posteromedial fragment in Mason and Molloy type 2B with one or more screws, or plate, if it is displaced more than 2 mm. Deltoid ligament injuries are repaired if incarcerated between medial malleolus and talus. The posteromedial fragment in Mason and Molloy type 2B will be fixed with one or more screws, or plate, if this fragment is displaced more than 2 mm. A Tillaux-Chaput or Wagstaffe fragment is fixed with suture anchor, plate, screw or pin if displaced >2 mm depending on size and comminution of the fragment.
  The syndesmosis is tested under fluoroscopy by lateralizing and then externally rotating the talus. If unstable it is fixed with one or two 3.5 mm cortical screws or a suture button.
  Interventions: Procedure: Fixation of the posterior malleolus fractures; Procedure: Fixation of lateral and/or medial malleolus fractures; Procedure: Syndesmotic fixation
- Non-fixation group (Active Comparator): Patients are placed in a supine position on the operating table. No fixation of the PMF. The PMF is reduced by ligamentotaxis. Lateral and/or medial malleolus fractures will be treated with ORIF if present.
  ORIF of the posteromedial fragment in Mason and Molloy type 2B with one or more screws, or plate, if it is displaced more than 2 mm.
  Deltoid ligament injuries are repaired if incarcerated between medial malleolus and talus.
  A Tillaux-Chaput or Wagstaffe fragment is fixed with suture anchor, plate, screw or pin if displaced >2 mm depending on size and comminution of the fragment.
  The syndesmosis is tested under fluoroscopy by lateralizing and then externally rotating the talus. If unstable it is fixed with one or two 3.5 mm cortical screws or a suturebutton.
  Interventions: Procedure: Fixation of lateral and/or medial malleolus fractures; Procedure: Syndesmotic fixation

INTERVENTIONS:
Procedure: Fixation of the posterior malleolus fractures — Fixation of the posterior malleolus fracture with screws and or plating.
  Arms: Fixation group
Procedure: Fixation of lateral and/or medial malleolus fractures — Fixation with screws and/or plating
Procedure: Syndesmotic fixation — Fixation of unstable syndesmosis with one or two 3.5 mm tricortical screws, or with a suture button.

SUMMARY:
Ankle fractures constitute 9% of all fractures and have an incidence of approximately 187 per 100,000 persons per year in Norway. A posterior malleolar fragment (PMF), located on the lower backside of the tibia, is present in up to 46% of Weber B. Weber B fractures are the most common type of fractures of the fibula, located at the height of the syndesmosis. Patients with a PMF were recently shown to have significantly lower patient-reported outcome measures (PROM) than the general population. For this reason, the indication and choice of intervention for these fractures have been the object of increased interest over the recent years. It is one of the most debated areas within ankle fracture surgery. Traditionally, these PMFs have been treated with closed reduction, without direct manipulation of the PMF, anteroposterior screw fixation, or even no-fixation of the smaller fragments. A more novel posterior approach to the ankle for open reduction and internal fixation is increasingly popular and has led to fixation of smaller and medium-sized PMFs. Studies suggest fracture reduction is better with a posterior approach. However, there is no consensus as to what the best treatment is. There are no available randomized controlled studies examining PROM in patients after surgery with fixation versus no fixation for the PMF.

Through a multicenter prospective randomized controlled trial initiated from Haukeland University Hospital, patients will be recruited and randomized to receive treatment with or without fixation of the PMF. Patients will be recruited at six study hospitals from all Regional Health Trusts in Norway. Treatment today is often based on local tradition and retrospective, ambiguous literature. As there is no clear evidence supporting the choice to fixate, or not fixate, the posterior malleolus fracture. The current study can contribute new knowledge and thereby contribute to an evidence-based approach to treating these patients.

Mason and Molly type 2A and 2B fractures will be included in the study.

DETAILED DESCRIPTION:
Ankle fractures constitute 9% of all fractures and have an incidence of approximately 187 per 100,000 persons per year in Norway. Weber B fractures are the most common type of fracture of the fibula. A posterior malleolar fragment (PMF) is present in up to 46% of Weber B and Weber C fractures. Patients with a PMF were recently shown to have significantly lower patient-reported outcome measures (PROM) than the general population. Clinical outcome for ankle fractures with a PMF is known to be poor from several studies. For this reason, the indication and choice of intervention for these fractures have been the object of increased interest over the recent years. It is one of the most debated areas within ankle fracture surgery. Traditionally, PMFs have been treated with closed reduction, without direct manipulation of the PMF, and anteroposterior screw fixation, or even no-fixation of the smaller fragments. A more novel posterior approach to the ankle for open reduction and internal fixation is increasingly popular and has led to fixation of smaller and medium-sized PMFs.

The reason for focusing on the posterior approach is new knowledge that intraarticular step-off in the tibiotalar joint and malreduced syndesmosis is associated with poor outcomes. Studies suggest fracture reduction is better with a posterior approach. However, there is no consensus as to what the best treatment is. Pilskog et. al. published a retrospective study in Nov. 2020 where patients without fixation reported similar PROM to patients with fixation. Most studies are retrospective and with a variable number of patients without a reasonable conclusion as to what is best practice. A few prospective studies are published. But there are no available randomized controlled studies examining PROM in patients after surgery with fixation versus no fixation for the PMF.

Through a multicenter, prospective, randomized controlled trial initiated from Haukeland University Hospital, patients with Weber B fracture and associated PMF (with or without a medial malleolus fracture) will be recruited and randomized to receive treatment with or without fixation of the PMF. Patients will be recruited at seven study hospitals from all Regional Health Trusts in Norway.

Mason and Molly type 2A and 2B fractures will be included in the study. Type 2 fractures are medium-sized fractures of the posterior malleolus which involve the fibular incisura. The fractures are classified as type 2A if only the posterior malleolus is fractured and as type 2B if there are two posterior fragments of the tibia in which the medial fragment extends to and involves the medial malleolus.

The lack of consensus on best practice is of great concern as patients of all ages are affected. In a retrospective study examining the patient-reported outcome of 130 patients with a PMF, 75% were aged 67 or younger. Such an injury, therefore, affects patients with many active years left in both their working life and daily activities. Interviews with the patient representative and with patients at the outpatient clinic reveal a long time for rehabilitation, over 16-18 months until 100% working ability. The patients also talk about the need to change working tasks due to reduced range of motion and pain. The study will not only answer the best way to treat the PMFs, but also give insights into the impact on the patient's life through the use of sick leave, treatment of the ankle syndesmosis, and complication rates. The aim is to give the patients the best possible treatment for better recovery and function.

The main aim of the study is to compare PROM in patients who had fixation of the PMF with patients without PMF fixation with the intention to define what is the best surgical approach and treatment of the fractures in question.

The null hypothesis (H0): There is no difference in mean patient-reported outcome (Self-reported Foot and Ankle Score, SEFAS) in patients treated with fixation of the PMF and patients treated without fixation of the PMF.

The intention is to deliver treatment recommendations based on the study results. The results will thus have direct consequences for both patients and orthopedic surgeons.

Additional aims:

* Publish treatment recommendations for ankle fractures including a PMF
* Sub-analysis of patients with and without syndesmotic injury
* Publish complication rates in the different treatment groups
* Health economic impact of ankle fractures
* Report rate of posttraumatic osteoarthritis after 2 and 5 years

The primary outcome is the summary score of Self-reported Foot and Ankle Score (SEFAS) at 2 years.

Project methodology:

Patients will be prospectively recruited from all six participating hospitals. An estimated 275 patients with ankle fractures per year will be eligible for inclusion. The investigators aim to include 208 patients over two years. Data are collected and stored by using Viedoc as the electronic case report form (eCRF). Patients will be treated according to randomization and data will be collected at each study site, stored via Viedoc, and sent to Haukeland University Hospital for analysis. Randomization is performed using Viedoc without interference from the surgeon on call. The last follow-up will be 5 years postoperative. Local coordinators at each hospital will manage inclusion and ensure correct treatment according to protocol.

The primary outcome of the mean difference between groups will be analyzed with an analysis of covariance (ANCOVA) with SEFAS at two years with baseline as covariate. Change in SEFAS over time (3 months - 1 year - 2 years - 5 years) will be analyzed with linear mixed effect models. The use of ANCOVA with adjusting for PROM at baseline (inclusion) is unique in orthopedic trauma studies as most studies report solely 1- or 2- year results with differences in mean values between groups. Adjusting for baseline will strengthen the analysis.

The Student t-test for continuous variables and chi-squared test for categorical variables will be used.

A power of 90% with a priori significance level of 0.05 requires 86 patients in each arm of randomization. A difference between groups of five points is considered to be a clinically relevant difference. Accounting for 20% lost to follow-up or dropout, 104 patients will be included in each group. The total number of patients will be 208.

NorCRIN will be used as a national monitoring service via Viedoc and Anne Mathilde Henden Kvamme.

Helse Bergen HF, Haukeland University Hospital, will be the coordinator of the project. All four regional health trusts in Norway are involved in this project. There will be responsible local coordinators for the study at the seven sites represented. The local coordinators are responsible for developing and coordinating the study and communicating with the project leaders and main coordinators.

Ethical considerations None of the surgical methods can be considered experimental as they are in conventional use at the study clinics and several other level 1 trauma centers. Participation in the study will not cause any delay in treatment compared to conventional care, nor will patients have any extra expenses related to follow-up evaluation. Patients having any concerns throughout the study period will be offered an extra follow-up by one of the participating surgeons.

As there is no clear evidence supporting the choice to fixate, or not fixate, the posterior malleolus fracture, the study can contribute new knowledge thereby contributing to a more evidence-based approach to treating these patients.

The project is approved by the Helse Bergen Data Protection Officer and Regional Committees for Medical and Health Research Ethics (REC). REC ref.nr: 255548. Patients will have to give their written, informed consent prior to inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

* Posterior malleolar (PM) fracture, of Mason & Molly type 2A/2B, associated with Weber B lateral malleolar fracture, with or without medial malleolar fracture
* Posterior malleoli >=2 mm displaced (on CT in axial, sagital or coronal plane)
* Patients informed, written consent
* Age 18-65 years
* For inclusion axial CT images are examined

  * Measurements are performed 5 millimeters (mm) cranial to the tibia plafond
  * Posterior malleolus fractures involving less than 40% of the fibular notch are included.

Exclusion Criteria:

* Non-compliant patient, i.e.: dementia, alcohol- or substance abuse
* ASA-4 patients
* Known congenital bone decease
* Pathological fractures
* Immunocompromised patients
* Tourists or patients on a short-term work/study permit
* Previous injury or condition of the ipsilateral ankle or ipsilateral lower extremity with a resulting dysfunction
* Poor controlled diabetes
* Patients with known arterial insufficiency
* Open fractures
* Severely traumatized patients (ISS>16)
* Patient declines to participate in study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Self-Reported Foot and Ankle Score | 2 years postoperatively
  Foot and ankle specific questionnaire with 12 questions with 5 levels. Total score from 0 (worst) to 48 (best).

SECONDARY OUTCOMES:
EQ-5D 5L | Baseline, 12 weeks, 1 year, 2 years and 5 years postoperatively
  Generic patient reported outcome questionnaire, Presentation of both change from baseline to 12 weeks, 1 year, 2, years and 5 years postoperatively. Presentation of both EQ-5D-5L frequencies and proportions reported by dimension and level, EQ-5D VAS, and EQ-5D index score.
VAS of stiffness (0-100) | 12 weeks, 1 year, 2 years and 5 years postoperatively
  Level of stiffness in the treated ankle from 0 (No stiffness) to 100 (No movement due to stiffness)
Osteoarthritis | 2 years and 5 years postoperatively
  Osteoarthritis on plain radiographs at 2- and 5-years postoperative graded by the Kellgren Lawrence classification
Dorsiflexion | 6 weeks, 12 weeks, 2 years postoperatively
  - Dorsiflexion measured by goniometer
  o With knee in flexion and the foot on the floor. The patient leans forward as far as possible without the heel lifting. The angle between the floor and the anterior boarder of the tibia is measured with a digital goniometer.
Change in Self-reported Foot and Ankle Score (SEFAS) | Baseline, 12 weeks, 1 year, and 5 years postoperatively
  Foot and ankle specific questionnaire with 12 questions with 5 levels. Total score from 0 (worst) to 48 (best).

OTHER OUTCOMES:
Anchor questions for evaluation of prom | Baseline (Generic health question). Alle questions: 3 months, 1 year, 2 years and 5 years postoperatively
  Generic and organ specific anchor questions for evaluation of SEFAS results and for patients satisfaction evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Jonas M Fevang, PhD, Study Director — Helse Bergen, Haukeland University Hospital; Jostein S Nilsen, MD, Principal Investigator — Helse Bergen, Haukeland University Hospital; Kristian Pilskog, MD, Principal Investigator — Helse Bergen, Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Orthopedic department, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bartonicek J, Rammelt S, Kostlivy K, Vanecek V, Klika D, Tresl I. Anatomy and classification of the posterior tibial fragment in ankle fractures. Arch Orthop Trauma Surg. 2015 Apr;135(4):505-16. doi: 10.1007/s00402-015-2171-4. Epub 2015 Feb 24. PMID 25708027
- [Background] Pilskog K, Gote TB, Odland HEJ, Fjeldsgaard KA, Dale H, Inderhaug E, Fevang JM. Traditional Approach vs Posterior Approach for Ankle Fractures Involving the Posterior Malleolus. Foot Ankle Int. 2021 Apr;42(4):389-399. doi: 10.1177/1071100720969431. Epub 2020 Nov 17. PMID 33203272
- [Background] Coster MC, Rosengren BE, Karlsson MK, Carlsson A. Age- and Gender-Specific Normative Values for the Self-Reported Foot and Ankle Score (SEFAS). Foot Ankle Int. 2018 Nov;39(11):1328-1334. doi: 10.1177/1071100718788499. Epub 2018 Jul 23. PMID 30035614
- [Background] Stufkens SA, van den Bekerom MP, Kerkhoffs GM, Hintermann B, van Dijk CN. Long-term outcome after 1822 operatively treated ankle fractures: a systematic review of the literature. Injury. 2011 Feb;42(2):119-27. doi: 10.1016/j.injury.2010.04.006. No abstract available. PMID 20444447
- [Background] Mason LW, Kaye A, Widnall J, Redfern J, Molloy A. Posterior Malleolar Ankle Fractures: An Effort at Improving Outcomes. JB JS Open Access. 2019 Jun 7;4(2):e0058. doi: 10.2106/JBJS.OA.18.00058. eCollection 2019 Apr-Jun. PMID 31334465
- [Background] Mingo-Robinet J, Lopez-Duran L, Galeote JE, Martinez-Cervell C. Ankle fractures with posterior malleolar fragment: management and results. J Foot Ankle Surg. 2011 Mar-Apr;50(2):141-5. doi: 10.1053/j.jfas.2010.12.013. PMID 21353996
- [Background] Hoogendoorn JM. Posterior Malleolar Open Reduction and Internal Fixation Through a Posterolateral Approach for Trimalleolar Fractures. JBJS Essent Surg Tech. 2017 Oct 25;7(4):e31. doi: 10.2106/JBJS.ST.17.00016. eCollection 2017 Dec 28. PMID 30233966
- [Background] Gandham S, Millward G, Molloy AP, Mason LW. Posterior malleolar fractures: A CT guided incision analysis. Foot (Edinb). 2020 Jun;43:101662. doi: 10.1016/j.foot.2019.101662. Epub 2019 Dec 30. PMID 32086138
- [Background] Tornetta P 3rd, Ricci W, Nork S, Collinge C, Steen B. The posterolateral approach to the tibia for displaced posterior malleolar injuries. J Orthop Trauma. 2011 Feb;25(2):123-6. doi: 10.1097/BOT.0b013e3181e47d29. PMID 21245717
- [Background] Verhage SM, Boot F, Schipper IB, Hoogendoorn JM. Open reduction and internal fixation of posterior malleolar fractures using the posterolateral approach. Bone Joint J. 2016 Jun;98-B(6):812-7. doi: 10.1302/0301-620X.98B6.36497. PMID 27235525
- [Background] Miller AN, Carroll EA, Parker RJ, Helfet DL, Lorich DG. Posterior malleolar stabilization of syndesmotic injuries is equivalent to screw fixation. Clin Orthop Relat Res. 2010 Apr;468(4):1129-35. doi: 10.1007/s11999-009-1111-4. Epub 2009 Oct 2. PMID 19798540
- [Background] Gardner MJ, Brodsky A, Briggs SM, Nielson JH, Lorich DG. Fixation of posterior malleolar fractures provides greater syndesmotic stability. Clin Orthop Relat Res. 2006 Jun;447:165-71. doi: 10.1097/01.blo.0000203489.21206.a9. PMID 16467626
- [Background] Tosun B, Selek O, Gok U, Ceylan H. Posterior Malleolus Fractures in Trimalleolar Ankle Fractures: Malleolus versus Transyndesmal Fixation. Indian J Orthop. 2018 May-Jun;52(3):309-314. doi: 10.4103/ortho.IJOrtho_308_16. PMID 29887634
- [Background] Hermans JJ, Beumer A, de Jong TA, Kleinrensink GJ. Anatomy of the distal tibiofibular syndesmosis in adults: a pictorial essay with a multimodality approach. J Anat. 2010 Dec;217(6):633-45. doi: 10.1111/j.1469-7580.2010.01302.x. PMID 21108526
- [Background] Jayatilaka MLT, Philpott MDG, Fisher A, Fisher L, Molloy A, Mason L. Anatomy of the Insertion of the Posterior Inferior Tibiofibular Ligament and the Posterior Malleolar Fracture. Foot Ankle Int. 2019 Nov;40(11):1319-1324. doi: 10.1177/1071100719865896. Epub 2019 Aug 8. PMID 31390895
- [Background] Forberger J, Sabandal PV, Dietrich M, Gralla J, Lattmann T, Platz A. Posterolateral approach to the displaced posterior malleolus: functional outcome and local morbidity. Foot Ankle Int. 2009 Apr;30(4):309-14. doi: 10.3113/FAI.2009.0309. PMID 19356354
- [Background] Ovaska MT, Makinen TJ, Madanat R, Kiljunen V, Lindahl J. A comprehensive analysis of patients with malreduced ankle fractures undergoing re-operation. Int Orthop. 2014 Jan;38(1):83-8. doi: 10.1007/s00264-013-2168-y. Epub 2013 Nov 20. PMID 24252973
- [Background] Amorosa LF, Brown GD, Greisberg J. A surgical approach to posterior pilon fractures. J Orthop Trauma. 2010 Mar;24(3):188-93. doi: 10.1097/BOT.0b013e3181b91927. PMID 20182256
- [Background] Weber M. Trimalleolar fractures with impaction of the posteromedial tibial plafond: implications for talar stability. Foot Ankle Int. 2004 Oct;25(10):716-27. doi: 10.1177/107110070402501005. PMID 15566703
- [Background] Little MT, Berkes MB, Lazaro LE, Sculco PK, Helfet DL, Lorich DG. Complications following treatment of supination external rotation ankle fractures through the posterolateral approach. Foot Ankle Int. 2013 Apr;34(4):523-9. doi: 10.1177/1071100713477626. Epub 2013 Feb 27. PMID 23447507
- [Background] Mason LW, Marlow WJ, Widnall J, Molloy AP. Pathoanatomy and Associated Injuries of Posterior Malleolus Fracture of the Ankle. Foot Ankle Int. 2017 Nov;38(11):1229-1235. doi: 10.1177/1071100717719533. Epub 2017 Jul 31. PMID 28758439
- [Background] Meijer DT, Doornberg JN, Sierevelt IN, Mallee WH, van Dijk CN, Kerkhoffs GM, Stufkens SA; Ankle Platform Study Collaborative - Science of Variation Group; Ankle Platform Study Collaborative - Science of Variation Group. Guesstimation of posterior malleolar fractures on lateral plain radiographs. Injury. 2015 Oct;46(10):2024-9. doi: 10.1016/j.injury.2015.07.019. Epub 2015 Jul 26. PMID 26253385
- [Background] Rammelt S, Bartonicek J, Neumann AP, Kroker L. [Fractures of the anterolateral tibial rim : The fourth malleolus]. Unfallchirurg. 2021 Mar;124(3):212-221. doi: 10.1007/s00113-021-00959-y. Epub 2021 Feb 12. German. PMID 33580301
- [Background] Rammelt S, Bartonicek J, Schepers T, Kroker L. Fixation of anterolateral distal tibial fractures: the anterior malleolus. Oper Orthop Traumatol. 2021 Apr;33(2):125-138. doi: 10.1007/s00064-021-00703-0. Epub 2021 Mar 22. PMID 33751133
- [Background] Fisher A, Bond A, Philpott MDG, Jayatilaka MLT, Lambert LA, Fisher L, Weigelt L, Myatt D, Molloy A, Mason L. The anatomy of the anterior inferior tibiofibular ligament and its relationship with the Wagstaffe fracture. Foot Ankle Surg. 2021 Apr;27(3):291-295. doi: 10.1016/j.fas.2021.01.003. Epub 2021 Jan 7. PMID 33446454
- [Background] B.G., Weber VHHB. Classification of ankle fractures. Die Verletzungen des oberen Sprung-gelenkes. 1972;(2nd ed.).
- [Background] Metsemakers WJ, Morgenstern M, McNally MA, Moriarty TF, McFadyen I, Scarborough M, Athanasou NA, Ochsner PE, Kuehl R, Raschke M, Borens O, Xie Z, Velkes S, Hungerer S, Kates SL, Zalavras C, Giannoudis PV, Richards RG, Verhofstad MHJ. Fracture-related infection: A consensus on definition from an international expert group. Injury. 2018 Mar;49(3):505-510. doi: 10.1016/j.injury.2017.08.040. Epub 2017 Aug 24. PMID 28867644
- [Background] McHale S, Williams M, Ball T. Retrospective cohort study of operatively treated ankle fractures involving the posterior malleolus. Foot Ankle Surg. 2020 Feb;26(2):138-145. doi: 10.1016/j.fas.2019.01.003. Epub 2019 Jan 18. PMID 30709682